CLINICAL TRIAL: NCT01079897
Title: A Randomized, Comparator-controlled, Double-blind, Multicenter Intra-individual Clinical Trial to Evaluate the Efficacy and Safety of an Ectoine-containing Cream in the Treatment of Mild to Moderate Atopic Dermatitis
Brief Title: Efficacy and Safety of an Ectoine-containing Cream in the Treatment of Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 133-002; 0010287 (Registry Identifier: DIMDI)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Mild to Moderate Atopic Dermatitis
Keywords: Atopic dermatitis; Ectoine; Treatment; Atopiclair; Medical device
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atopiclair (Active Comparator)
  Interventions: Device: Atopiclair
- EHK02-01 (Experimental): Ectoine containing cream
  Interventions: Device: EHK02-01

INTERVENTIONS:
Device: Atopiclair — topical applied cream, twice daily
  Other Names: Zarzenda; MAS063DP; Atopiclair non-steroidal cream
  Arms: Atopiclair
Device: EHK02-01 — topical applied cream containing 7% ectoine
  Other Names: ectoine-containing cream,; 7% Ectoin
  Arms: EHK02-01

SUMMARY:
This study evaluates the efficacy of the topical used ectoine-formulation EHK02-01 compared to Atopiclair. Patients are examined at visit 2 (baseline visit). The patient topically applies EHK02-01 or Zarzenda® twice daily on two symmetric lesional areas over 28 days. Response to therapy is recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Female or male individuals between 18 and 65 years in good general health diagnosed atopic dermatitis for ≥ 6 months, in active stage (active stage means severity as measured by overall IGA-Score between 1 and 4)
* At least two comparable areas of stable atopic eczema on bilateral symmetric corresponding sides of the extremities or the body (except for head and genital area), each of at least 10 cm², with a modified, objective local SCORAD of the test areas > 5
* Both lesional areas of interest must have a difference in the modified, objective local SCORAD of ≤ 3
* Willingness to adhere to the schedule of the investigation, concomitant therapy prohibitions, restrictions, treatment regimen and procedures described in the CIP
* Written informed consent to participate in the trial, prior to any investigation related procedures, indicating an understanding of the purpose of the clinical investigation
* A patient of childbearing potential agrees to use a contraceptive methods for the duration of the investigation according to CPMP/ICH 286/95 note 3

Exclusion Criteria:

* Patients who are self-reported to be pregnant, nursing or planning pregnancy during the clinical investigation
* Patients with any skin disease that in the investigator's opinion may interfere with the conduct of the study or the evaluation of the results (e.g. psoriasis)
* Patients with a known malignancy
* Presence of any disease and/or condition and/or history of diseases and/or conditions that according to the investigator may interfere with the conduct of the investigation or the evaluation of the results (such as abnormal laboratory values, chronic inflammatory dis-eases, immunosuppressive diseases, autoimmune diseases, liver or kidney diseases, severe infectious diseases)
* Patients who did not respect the wash-out periods prior to and during the clinical investigation
* Vaccination within 6 days prior to enrolment and during the study.
* Patients with a known allergy against any ingredient of the test products
* Patients who are known to have had a substance abuse (drug or alcohol) problem within the previous 12 months
* Patients who participate in another clinical trial or have participated in another clinical trial within the last 30 days prior to the first day of investigation
* Patients who are involved in the organization of the clinical investigation
* Patients that are in any way dependant on the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
change of a modified, objective (local) SCORAD | 28 days

SECONDARY OUTCOMES:
Change of local IGA | 28 days
Change of Pruritus | 28 days
Patient's judgment on efficacy | 28 days
AEs during treatment phase | 28 days
Physical examination | 28 days
Patient's assessment of tolerability and safe | 28 days
change of the modified, objective local SCORAD | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Vanscheidt, Professor, Principal Investigator — Professor Dr. med Wolfgang Vanscheid (Hautarzt, Allergologie, Phlebologie); Tanja Fischer, Dr., Principal Investigator — Haut- und Lasercentrum Potsdam; Martin Miehe, Dr., Principal Investigator — Hautarztzentrum Tegel; Michael Sebastian, Dr., Principal Investigator — Facharzt für Dermatologie
Locations (4):
- Germany (4):
  - Hautarztzentrum Tegel, Berlin
  - Hautarztpraxis, Freiburg im Breisgau
  - Gemeinschaftspraxis Mahlow, Mahlow
  - Haut- und Lasercentrum Potsdam, Potsdam